CLINICAL TRIAL: NCT00171093
Title: A 10-12 Week Multicenter, Double-blind Study to Evaluate the Efficacy and Safety of the Combination of Valsartan (320 mg) and Simvastatin (80 mg) Compared to Valsartan (320 mg) and Simvastatin (80 mg) Monotherapies in Essential Hypertension and Hypercholesterolemia
Brief Title: A 10-12 Week Study to Evaluate the Safety and Efficacy of 320 mg Valsartan and 80 mg Simvastatin in Combination and as Monotherapies in Treating Hypertension and Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAS489A2316
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: HYPERTENSION; HYPERCHOLESTEROLEMIA
Keywords: HYPERTENSION; HYPERCHOLESTEROLEMIA; BLOOD PRESSURE; CHOLESTEROL; VALSARTAN; SIMVASTATIN
MeSH Terms: conditions — Hypertension; Hypercholesterolemia | interventions — Valsartan; Simvastatin

INTERVENTIONS:
Drug: valsartan + simvastatin

SUMMARY:
This 10-12 week study will provide data on the safety and efficacy of using 320 valsartan and 80 mg simvastatin together compared to using either one alone in lowering blood pressure and LDL cholesterol. After discontinuing current drug therapies for hypertension and hypercholesterolemia, patients will be given 320mg valsartan+80mg simvastatin, 320mg valsartan+placebo, or 80mg simvastatin+placebo..

ELIGIBILITY:
Inclusion Criteria:

* ESSENTIAL HYPERTENSION
* ELEVATED LDL-C CHOLESTEROL
* USING STABLE DOSE OF HMG CoA REDUCTASE INHIBITOR (STATIN) FOR 3+ MONTHS

Exclusion Criteria:

* SEVERE HYPERTENSION
* EVIDENCE OF HISTORY OR CURRENT HEART DISEASE
* HISTORY OF STROKE OR MYOCARDIAL INFARCTION
* DISLIPIDEMIA OR HYPERTENSION DUE TO SECONDARY CAUSES
* UNCONTROLLED DIABETES OR INSULIN

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 369
Dates: Start 2004-09; Primary Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Change in average ambulatory systolic blood pressure over 24 hours
Change in serum low density lipoprotein cholesterol (LDL-C )

SECONDARY OUTCOMES:
Adverse events and serious adverse events at each study visit for 42 days
Change in average ambulatory systolic blood pressure over 24 hours between two different treatment therapies
Change in 24 hour ambulatory blood pressure in the daytime compared to nighttime
Change in 24 hour ambulatory blood pressure 21-24 hours after last dose of study medication
Change in total cholesterol, triglycerides, and high densitiy lipoprotein cholesterol (HDL-C) from baseline after 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States